CLINICAL TRIAL: NCT06351215
Title: Use of Single-Dose Oral Methadone for Pain Management in Outpatient Arthroscopic Hip and Knee Procedures
Brief Title: PO Methadone Ortho Outpatient
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Keck School of Medicine of USC (Other)
Responsible Party: Principal Investigator, Abigail Song, Co-Investigator, Keck School of Medicine of USC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APP-24-00554
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Arthroscopic Knee Repair; Arthroscopic Hip Repair
Keywords: arthroscopic knee repair; arthroscopic hip repair; oral methadone; post-operative pain control; ambulatory surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): placebo sugar pill and standard intraoperative pain control using short-acting opioids, with drug choice and dosing at the practitioner's discretion
  Interventions: Drug: Placebo
- Interventional (Experimental): 5mg PO methadone for participants <50kg or 10mg PO methadone for participants >50kg
  Interventions: Drug: Methadone group

INTERVENTIONS:
Drug: Methadone group — 5mg PO methadone for participants <50kg or 10mg PO methadone for participants >50kg
  Arms: Interventional
Drug: Placebo — sugar pill that is identical look-alike to study drug
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if oral methadone given before surgery works to minimize post-operative pain and opioid usage. The main questions it aims to answer are:

Does oral methadone improve post-operative pain scores as compared to standard treatment? Does oral methadone lead to reduced use of post-operative and post-discharge opioid usage as compared to the current standard treatment?

Researchers will compare oral methadone to a placebo (a look-alike substance that contains no drug) to assess the questions above.

Participants will:

Receive either oral methadone or a look-alike placebo before surgery Receive standard intraoperative and immediate post-operative pain control at the anesthesiologist's discretion Be asked about their pain levels in the recovery area Keep a diary of pain and opioid usage over the first 2 days after surgery

DETAILED DESCRIPTION:
STUDY METHOD We plan to perform a double-blinded randomized control study, where the participants, anesthesiologist, data collectors, and study team will be unaware of the intervention offered. Participants will be randomly assigned to the control group (standard intraoperative pain control using short-acting opioids, with drug choice and dosing at the practitioner's discretion) or to the intervention group (a single dose of perioperative oral methadone).

Patients will be recruited and consented to whether they want to participate in the study by a member of the team during a pre-operative clinic visit (Anesthesia START clinic or orthopedic surgery clinic) or on day-of-surgery in the pre-op holding area.

Participants will be randomized to either the control group or treatment group using randomization software. Participants assigned to the intervention group will receive a single dose of oral methadone will be administered in the pre-operative holding area. Dosing will be weight dependent, using 0.15mg/kg ideal body weight (IBW) as a reference; participants weighing less than 50kg will receive 5mg oral methadone, while participants weighing more than 50kg will receive 10mg oral methadone. Participants assigned to the control group will receive an identical-looking placebo sugar pill. A study pharmacist will deliver the appropriate pill to the patient or pre-op nurse in the pre-op holding area on the day of surgery.

Pre-operatively, all participants will complete a survey collecting data on visual analog scale (VAS) pain scores for the 2 weeks leading up to surgery, whether this is different from their baseline pain score at home (if applicable), and pre-operative opioid usage (if applicable). All participants will receive standard-of-care pre-operative non-opioid medications as determined by the orthopedic surgical team if needed.

Intraoperatively, participants will receive either GA or monitored anesthesia care, at the discretion of the anesthesia care team.

In the post-anesthesia acute care unit (PACU), all participants will receive standard PACU medications (ie. intravenous dilaudid or oral oxycodone, and acetaminophen as needed) for pain relief. Pain scores on a 1-10 scale and amount of opioid usage will be collected per standard PACU protocol upon arrival, after 30 minutes, and after 60 minutes. Post-discharge, all participants will receive oxycodone-acetaminophen for at-home pain (as standardized by the orthopedic surgery team) to be used as needed for breakthrough pain refractory to acetaminophen/ibuprofen, or in patients where these medications are contraindicated.

Following discharge, a member of the study team will call participants on post-operative day 1 and post-operative day 2 to assess pain scores and opioid usage. Participants will also be discharged with a pain diary to assist in documenting endpoints. They will also be asked to document any complications or adverse events at each of these time intervals.

Once the data collection is complete, we will perform statistics (detailed below) to determine if there is any significant difference. The primary outcome will be post-discharge opioid usage, and the secondary outcome will be patient-perceived pain scores at the time intervals above.

STRATIFICATION/DESCRIPTIVE FACTORS/RANDOMIZATION SCHEME

Participants will not be stratified prior to randomization.

Descriptive factors: age, gender, BMI will be looked to assess for possible confounding variables, but will not affect group assignment.

The website randomizer.org will assist in our randomization of participants enrolled in the study. The software randomly determines which participant will be assigned to Control vs Treatment group in a 1:1 ratio. At the onset of the study, we will create a predetermined randomization list (containing study participant code and treatment arm assignment), and provide it to the study pharmacist who will then be the only one with access to this linked info. The study pharmacist will be informed of the new enrollment and will read back the study code to the team member, who will record it in a separate data collection form that contains link between Medical Record Number and participant code. The pharmacist will strike out the participant code on their sheet to keep track of used codes, then prepare the appropriate medication and deliver it to the participant or pre-op nurse in the pre-op holding area on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* medically optimized participants who will undergo elective arthroscopic knee or hip repair

Exclusion Criteria:

* pregnant or breastfeeding, age under 18, history of respiratory compromise, allergy to opioids, recipient of pre-operative nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Post-op opioid usage | at Post-Anesthesia Care Unit arrival, post-operative 30 minutes, post-op 60 minutes, post-operative day 1, and post-operative day 2
  opioid usage, as measured in morphine equivalent doses (MED)

SECONDARY OUTCOMES:
Post-op Pain Score | at Post-Anesthesia Care Unit arrival, post-operative 30 minutes, post-op 60 minutes, post-operative day 1, and post-operative day 2
  pain scores on the visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, M.D., Principal Investigator — Keck School of Medicine of USC
Locations (1):
- USC Healthcare Consultation 3, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Vender JS, Benson J, Newmark RL. Clinical Effectiveness and Safety of Intraoperative Methadone in Patients Undergoing Posterior Spinal Fusion Surgery: A Randomized, Double-blinded, Controlled Trial. Anesthesiology. 2017 May;126(5):822-833. doi: 10.1097/ALN.0000000000001609. PMID 28418966
- [Background] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Background] Murphy GS, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Dickerson D, Bilimoria S, Benson J, Maher CE, Trenk GJ, Teister KJ, Szokol JW. Postoperative Pain and Analgesic Requirements in the First Year after Intraoperative Methadone for Complex Spine and Cardiac Surgery. Anesthesiology. 2020 Feb;132(2):330-342. doi: 10.1097/ALN.0000000000003025. PMID 31939849
- [Background] Murphy GS, Avram MJ, Greenberg SB, Benson J, Bilimoria S, Maher CE, Teister K, Szokol JW. Perioperative Methadone and Ketamine for Postoperative Pain Control in Spinal Surgical Patients: A Randomized, Double-blind, Placebo-controlled Trial. Anesthesiology. 2021 May 1;134(5):697-708. doi: 10.1097/ALN.0000000000003743. PMID 33730151
- [Background] Komen H, Brunt LM, Deych E, Blood J, Kharasch ED. Intraoperative Methadone in Same-Day Ambulatory Surgery: A Randomized, Double-Blinded, Dose-Finding Pilot Study. Anesth Analg. 2019 Apr;128(4):802-810. doi: 10.1213/ANE.0000000000003464. PMID 29847382
- [Background] Kharasch ED, Brunt LM, Blood J, Komen H. Intraoperative Methadone in Next-day Discharge Outpatient Surgery: A Randomized, Double-blinded, Dose-finding Pilot Study. Anesthesiology. 2023 Oct 1;139(4):405-419. doi: 10.1097/ALN.0000000000004663. PMID 37350677
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] undefined